CLINICAL TRIAL: NCT06458296
Title: Evaluating the Efficacy of AI-Guided vs. Standard Physician-Guided Dietary Supplement Prescriptions for Weight Loss in Obese Patients: A Randomized Controlled Pilot Trial
Brief Title: Evaluating the Efficacy of AI-Guided (GenAIS TM) vs. Standard Physician-Guided Dietary Supplement Prescriptions for Weight Loss in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Collaborators: Center of New Medical Technologies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SW013
Record Dates: First submitted 2024-06-04; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Obesity
Keywords: Dietary Supplements; AI-guided prescriptions; Genetic profiling; Metabolic profiling
MeSH Terms: conditions — Obesity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator)
  Interventions: Other: Control Group
- AI-Guided Group (Experimental)
  Interventions: Other: AI-Guided Group

INTERVENTIONS:
Other: Control Group — Participants receive DS prescriptions from a physician based on current standard practices, which include biochemical markers, genetic data, and metabolic profiles.
  Arms: Control Group
Other: AI-Guided Group — Participants receive DS prescriptions determined by an AI system, which considers genetic data, metabolic profiles, biochemical markers, and patient history.
  Arms: AI-Guided Group

SUMMARY:
Obesity, a chronic disease characterized by excessive fat accumulation, significantly impacts health. Genetic factors influence the development of obesity by affecting behavioral, dietary habits, and metabolic processes. This study investigated whether dietary supplements (DS), personalized through genetic and metabolic profiling, could enhance weight loss when combined with physical activity and dietary changes. The objective was to compare the efficacy of standard physician-guided DS prescriptions with AI-guided DS prescriptions in promoting weight loss in obese patients. The hypothesis was that AI-guided DS prescriptions, utilizing detailed genetic and metabolic data, would be more effective in promoting weight loss than standard physician-guided DS prescriptions. This was a 6-month randomized, controlled pilot clinical trial with an additional 6-month follow-up. Participants were healthy individuals aged 40-60 years with a BMI of 25 or greater. Participants were excluded if they had significant medical conditions or recent changes in medication or supplements. They were randomly assigned to either the control group (physician-guided DS prescriptions) or the AI-guided group (AI-determined DS prescriptions). The AI system developed by Triangel Scientific analyzed genetic, metabolic, and biochemical data to personalize treatment. Baseline measurements included comprehensive metabolic panels, genetic testing, metabolomic profiling, and detailed patient history

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants aged between 40 and 60 years.
* BMI of 25 or greater and no more than a 3% change in body mass within the last three months.

Exclusion Criteria:

* Individuals who have taken any prescribed medications or dietary supplements in the two weeks prior to the study.

  * Those with a clinically significant history of major digestive, liver, kidney, cardiovascular, hematological diseases, diabetes, gastrointestinal disorders, or any other serious acute or chronic medical conditions.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
percentage change in body weigh | 180 days

SECONDARY OUTCOMES:
Change in BMI | 180 days
Percent change in high-sensitivity C-reactive | 180 days
Percent change in fasting glucose | 180 days
Percent change in insulin | 180 days
Percent change in total cholesterol | 180 days
Percent change in Low density lipoproteids | 180 days
Percent change in high density lipoprodeids | 180 days
Percent change in triglycerides | 180 days
Appetite ratings using visual analogue scale change | 180 days
  The scale has minimum of 0 - no appetite and 10 as a good appetite

CONTACTS AND LOCATIONS:
Locations (1):
- Center of New Medical Technologies, Novosibirsk, Novosibisk Region, Russia

REFERENCES:
- [Derived] Pokushalov E, Garcia C, Ponomarenko A, Samoilova I, Smith J, Johnson M, Pak I, Shrainer E, Kudlay D, Romanova A, Miller R. Optimizing weight loss with artificial intelligence: A randomized controlled trial of dietary-supplement prescriptions in adults with overweight and obesity. Clin Nutr ESPEN. 2025 Oct;69:75-86. doi: 10.1016/j.clnesp.2025.06.035. Epub 2025 Jun 23. PMID 40562096